CLINICAL TRIAL: NCT04527679
Title: Combined Therapy Using Cisplatin and Gemcitabine Chemotherapy and Lenvatinib for Patients With Unresectable Intrahepatic Cholangiocarcinoma, a Single-arm Study
Brief Title: Cisplatin and Gemcitabine Chemotherapy and Lenvatinib for Patients With Unresectable Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zs-icc-len
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: intrahepatic Cholangiocarcinoma; Lenvatinib; GC chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC combined Lenvatinib (Experimental): 1. GC chemotherapy D1 Cisplatin 25mg/m2+ gemcitabine 1g/m2, D8 gemcitabine 1g/m2 Three weeks is a course of treatment, a total of 8 courses.
  2. Lenvatinib (<60kg: 8mg /d; ≥60kg, 12mg).
  Interventions: Drug: GC combined Lenvatinib

INTERVENTIONS:
Drug: GC combined Lenvatinib — 1. GC chemotherapy D1 Cisplatin 25mg/m2+ gemcitabine 1g/m2, D8 gemcitabine 1g/m2 Three weeks is a course of treatment, a total of 8 courses.
  2. Lenvatinib (<60kg: 8mg /d; ≥60kg, 12mg).

SUMMARY:
We aim to explore the effects and safety of GC (Cisplatin and gemcitabine) chemotherapy combined with Lenvatinib as first-line therapy in advanced or unresectable intrahepatic cholangiocarcinoma

DETAILED DESCRIPTION:
For advanced intrahepatic cholangiocarcinoma (ICC) that cannot be surgically removed or accompanied by metastasis, the NCCN guidelines (NCCN guidelines hepatobiliary cancer, 2019) recommend that the current treatment options are limited, mainly recommending gemcitabine combined with platinum based antitumor drugs (cisplatin, oxaliplatin, etc.) chemotherapy as first-line treatment. Adding targeted drugs can enhance the anti-tumor effect. GC chemotherapy (Cisplatin + gemcitabine) has been used in the treatment of advanced intrahepatic cholangiocarcinoma, but the efficacy is still not satisfactory. Lenvatinib is a small-molecule multikinase inhibitor that is currently approved for first-line treatment of advanced hepatocellular carcinoma. Lenvatinib combined with chemotherapy may have a better effect than single use for advanced ICC. At present, lenvatinib combined with GC chemotherapy in the first-line treatment of advanced ICC has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must sign an informed consent form; 2. Age 18-75 years old, both male and female; 3. ECOG performance status score (PS score) 0 or 1; 4. Child-Pugh score A period; 5. Intrahepatic cholangiocarcinoma confirmed by histopathology; agree to provide previously-stored tumor tissue specimens or fresh biopsy tumor lesions; 6. Unresectable ICC patients or postoperative diagnosis of ICC recurrence and metastasis, have not received systemic treatment within 6 months; 7. The functional indicators of important organs meet the following requirements Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; T3, T4≤2 times the upper limit of normal value; Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; Serum creatinine ≤ 1.5 times the upper limit of normal value, creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula); 8. The subject has at least 1 measurable lesion (according to RECIST1.1); 9. For women who are not breastfeeding or pregnant, contraceptives during treatment or 3 months after the end of treatment.

Exclusion Criteria:

* 1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma and other non-biliary cell carcinoma malignant tumor components; 2. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma; 3. Have used Lenvatinib or gemcitabine-based chemotherapy within 6 months; 4. Severe cardiopulmonary and renal dysfunction; 5. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements); 6. Abnormal coagulation function (PT>14s), have a bleeding tendency or are receiving thrombolysis or anticoagulation therapy; 7. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000; 8. History of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment; 9. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period; 10. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive; 11. A history of psychotropic drug abuse, alcohol or drug abuse; 12. Known to have a history of severe allergies to any targeted anti-angiogenesis drugs, platinum or gemcitabine; 13. Other factors judged by the investigator that may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, severe laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  Objective response rate of advanced and unresectable intrahepatic cholangiocarcinoma

SECONDARY OUTCOMES:
Safety: the potential side effects | 12 months
  The potential side effects
Overall survival | 12 months
  From the beginning date of combined therapy to the date of death
Progression free survival | 12 months
  From the beginning date of combined therapy to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyong Huang, MD & PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Choi SB, Kim KS, Choi JY, Park SW, Choi JS, Lee WJ, Chung JB. The prognosis and survival outcome of intrahepatic cholangiocarcinoma following surgical resection: association of lymph node metastasis and lymph node dissection with survival. Ann Surg Oncol. 2009 Nov;16(11):3048-56. doi: 10.1245/s10434-009-0631-1. Epub 2009 Jul 22. PMID 19626372